CLINICAL TRIAL: NCT03391713
Title: The Effectiveness of Waiting Room Posters in Improving Awareness and Knowledge of the Signs and Symptoms of Stroke
Brief Title: The Effectiveness of Waiting Room Posters for Stroke Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Professor Su May Liew, Associate Professor, University of Malaya
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RU009-2017J
Record Dates: First submitted 2017-12-20; First posted 2018-01-05 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Stroke, Acute
Keywords: awareness; poster; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No exposure to waiting room posters
- Intervention (Active Comparator): During the second half of the study (two weeks), there will be an education poster in the waiting room of the clinic, fashioned after the Face, Arms, Speech, Time (FAST) poster developed by the American Heart Association (AHA), but in Malay.
  Interventions: Behavioral: Poster

INTERVENTIONS:
Behavioral: Poster — The poster includes the FAST symptoms but translated to the Malay language (Ce.P.A.T) Cakap tak jelas (slurred speech - Speech slurring) Perubahan muka (face changes - Face drooping) Anggota lemah (weak limbs - Arm weakness) Terus ke Hospital (straight to the hospital - Time to call 911
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine the effectiveness of posters in improving patient awareness and knowledge of the signs and symptoms of stroke. The control group study will be conducted in the first two weeks. Subsequently, the intervention arm will occur in the subsequent two weeks.

DETAILED DESCRIPTION:
Stroke is a major health problem and a known cause of death and disability worldwide. In Malaysia, stroke is known to be top five causes of death and top ten causes of hospitalization Malaysia. Ischemic stroke accounts for more than 95% of all stroke cases (1). A recent study done in Malaysia showed that only 26% of patients with stroke symptoms presented to the hospital within 3 hours. One of the reasons was patients did not perceive the symptoms of stroke as being that of a serious illness (2). One of the modalities to raise awareness of stroke is through an educational poster. Posters in the waiting room can increase awareness of health promotion issues (3). Therefore, by placing poster regarding sign and symptoms of stroke in the waiting room in a government clinic, can increase awareness of early presentation of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adult age more than 18 years old and above
* Able to understand Malay
* Able to provide informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1064 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Awareness of the signs and symptoms of stroke | Within 24 hours
  Participants awareness of the signs and symptoms of stroke as assessed by a questionnaire. For the symptoms, patients are scored from 0-7, according to each correct answer given.
  For the action taken, and the time frame, a score of either 0 or 1 is given, 1 being the right answer given.
  A higher score would indicate a better awareness of the signs and symptoms of stroke.

SECONDARY OUTCOMES:
Improvement in the knowledge of the need for a quick transfer to the hospital | Within 24 hours
  Knowledge of the need for a quick transfer to the hospital as assessed by a questionnaire. For the symptoms, patients are scored from 0-7, according to each correct answer given.
  For the action taken, and the time frame, a score of either 0 or 1 is given, 1 being the right answer given.
  A higher score would indicate a better awareness of the signs and symptoms of stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Su May Liew, Principal Investigator — University of Malaya
Locations (1):
- Klinik Kesihatan Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheah WK, Hor CP, Zariah AA, Looi I. A Review of Stroke Research in Malaysia from 2000 - 2014. Med J Malaysia. 2016 Jun;71(Suppl 1):58-69. PMID 27801388
- [Background] Factors associated with delay in seeking treatment by patients with acute stroke: The National Neurology Registry (NNeuR) of Malaysia . Malinee Neelamegam1, Sharad Malavade1, Irene Looi2, Norsima Nazifah Sidek3, Zariah Abdul Aziz3. 2014
- [Background] Ward K, Hawthorne K. Do patients read health promotion posters in the waiting room? A study in one general practice. Br J Gen Pract. 1994 Dec;44(389):583-5. PMID 7748670